CLINICAL TRIAL: NCT00001630
Title: High-Dose Cyclophosphamide With CD34+ Selected Autologous Hematopoietic Cell Support for Treatment of Refractory Chronic Autoimmune Thrombocytopenia
Brief Title: Treatment of Autoimmune Thrombocytopenia (AITP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 970154; 97-H-0154
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-21

CONDITIONS: Autoimmune Disease; Autoimmune Hemolytic Anemia; Thrombocytopenia
Keywords: Immunosuppression; Thrombocytopenia; Autoimmune Disease; Evan's Syndrome; Autoimmune Hemolytic Anemia; Episodic Bleeding
MeSH Terms: conditions — Autoimmune Diseases; Anemia, Hemolytic, Autoimmune; Thrombocytopenia; Evans Syndrome

INTERVENTIONS:
Device: Isolex 300i

SUMMARY:
Platelets are particles found along with red and white blood cells in the blood that play a role in the process of blood clotting. Disorders affecting the platelets can lower the amount of platelets in the blood and put patients at risk of bleeding. The condition of low platelets is referred to as thrombocytopenia.

Thrombocytopenia can be associated with a variety of diseases including cancer, leukemia, tuberculosis, or as a result of an autoimmune reaction. Autoimmune reactions are disorders in which the normal immune system begins attacking itself. Autoimmune thrombocytopenia (AITP) is a disorder of low blood platelet counts in which platelets are destroyed by antibodies produced by the immune system.

Unfortunately, many patients with AITP do not respond to standard treatments for thrombocytopenia. Cyclophosphamide is a drug that works to suppress the activity of the immune system. Researchers believe that combining this drug with transplanted rescued blood stem cells may provide effective treatment for AITP.

The purpose of this study is to explore the affordability and safety of this therapy for the treatment of AITP. The effectiveness of the therapy will be measured by the number of patients whose platelet levels rise greater than 100,000/m3.

If this treatment approach appears affordable, this study will form the basis for a larger study to compare alternate treatment approaches.

DETAILED DESCRIPTION:
Autoimmune Thrombocytopenia (AITP) is a disorder of low blood platelet counts in which platelet destruction is caused by antiplatelet autoantibodies. A large proportion of patients with chronic AITP are refractory to standard therapies including corticosteroids, immune globulin and splenectomy. Cyclophosphamide is a cytotoxic immunosuppressive agent which may induce durable remissions of refractory autoimmune diseases. High-dose cyclophosphamide with peripheral blood stem cell (PBPC) rescue has been proposed as a potential definitive therapy for AITP; however, the infusion of autoreactive lymphocytes could result in relapse. The use of PBPC depleted of T-lymphocytes could circumvent this limitation.

The purpose of this phase I/II study is to explore the feasibility and safety of this approach, and to seek preliminary evidence of effectiveness, of using high-dose cyclophosphamide (50 mg/kg/day x 4) followed by infusion of autologous PBPC enriched for CD34+ cells (concomitantly depleted of CD3+ cells) for the treatment of patients with refractory AITP. Safety/feasibility parameters to be examined will include the ability to mobilize, harvest and purify sufficient PBPC to yield greater than 2 x 10(6) CD34+ cells/kg; symptomatic acceptability and hematologic toxicities of the mobilization regimen (filgrastim 10 micrograms/kg/day IV); tolerability of the leukapheresis procedure, including the central line placement and maintenance; depth and duration of blood cell nadirs following chemotherapy; peritransplant bleeding episodes and transfusion requirements; episodes of febrile neutropenia, culture-proven infections and antibiotic usage. Effectiveness will be gauged by the rapidity and number of patients to achieve complete remission (platelet count greater than 100,000/mm(3) and partial remission (platelet count greater than 50,000/mm(3) or doubling of the platelet count with resolution of bleeding episodes). Ancillary evidence of therapeutic effect will be sought by examining changes in titers of platelet surface glycoprotein antibodies. In addition, alterations in T-lymphocyte subsets will be examined by flow cytometry. If this treatment approach appears feasible, this study will form the basis for a larger trial to compare alternate treatment approaches.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male or female, ages 18-65 years old.

Refractory severe chronic autoimmune thrombocytopenia, with or without autoimmune hemolytic anemia (Evan's syndrome), with all the following:

1. Platelet count frequently below 20,000/mm(3) despite active

   treatment for a period of greater than 6 months.
2. Normal or increased megakaryocytes on bone marrow

   aspirate/bx.
3. No plausible alternative etiology such as drug-mediated

   thrombocytopenia, marrow failure syndrome or thrombocytopenia

   related to viral or bacterial infection.
4. Failure of treatment with:

i. conventional-dose steroids (e.g., prednisone or dosage of 40

mg/day or equivalent, followed by dosage taper) for at least 3

months.

ii. intravenous immunoglobulin.

iii. splenectomy.

e. Episodic bleeding requiring transfusions or ecchymoses interfering

with ordinary daily activities.

EXCLUSION CRITERIA:

ECOG performance status greater than 1.

Cardiopulmonary disease including:

1. History of coronary artery disease, angina pectoris or congestive heart failure.
2. LV ejection fraction less than 40 percent by 2D echocardiogram.

Renal disease, serum creatinine greater than 2.5 mg/dL or creatinine clearance less than 30 mL/min.

Significant hepatic dysfunction, bilirubin greater than 2 mg/dL or transaminases greater than 2 times UNL.

Uncorrected coagulopathy.

Bone marrow aplasia (cellularity less than 10 percent), single or multilineage hematopoietic failure, myelodysplastic syndrome, or extensive marrow fibrosis.

History or active diagnosis of malignancy (except treated non-melanoma skin cancer or cevical carcinoma in situ).

HIV positive.

Pregnancy or lactation, unwillingness to practice adequate birth control in the peritransplant period.

Psychiatric illness or mental incapacity to understand and give informed consent.

Other medical illness or condition which, in the opinion of the Investigators, may contraindicate participation in this study due to patients' risk or compromise of study integrity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1997-07-21; Study Completion 2009-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Semple JW, Freedman J. Abnormal cellular immune mechanisms associated with autoimmune thrombocytopenia. Transfus Med Rev. 1995 Oct;9(4):327-38. doi: 10.1016/s0887-7963(05)80080-x. No abstract available. PMID 8541715
- [Background] Karpatkin S. Autoimmune (idiopathic) thrombocytopenic purpura. Lancet. 1997 May 24;349(9064):1531-6. doi: 10.1016/S0140-6736(96)12118-8. No abstract available. PMID 9167472
- [Background] George JN, el-Harake MA, Raskob GE. Chronic idiopathic thrombocytopenic purpura. N Engl J Med. 1994 Nov 3;331(18):1207-11. doi: 10.1056/NEJM199411033311807. No abstract available. PMID 7935660